CLINICAL TRIAL: NCT00020839
Title: Temozolomide Versus Temozolomide + Whole Brain Radiation In Stage IV Melanoma Patients With Asymptomatic Brain Metastases
Brief Title: Temozolomide With or Without Radiation Therapy to the Brain in Treating Patients With Stage IV Melanoma That Is Metastatic to the Brain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-18981; EORTC-18981
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Melanoma (Skin); Metastatic Cancer
Keywords: stage IV melanoma; recurrent melanoma; tumors metastatic to brain
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis; Brain Neoplasms | interventions — Temozolomide; Radiotherapy

INTERVENTIONS:
Drug: temozolomide
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known if chemotherapy is more effective with or without radiation therapy in treating brain metastases.

PURPOSE: Randomized phase III trial to compare the effectiveness of chemotherapy with or without radiation therapy to the brain in treating patients who have stage IV melanoma with asymptomatic brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of temozolomide with or without radiotherapy in terms of overall survival in patients with stage IV melanoma with asymptomatic brain metastases.
* Compare the time to appearance of neurological symptoms in patients treated with these regimens.
* Compare the progression-free survival of patients treated with these regimens.
* Compare the quality of life and quality-adjusted survival of patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to LDH levels (less than 225 U/L vs 225 U/L or more), concurrent metastases (visceral vs soft tissue), and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral temozolomide once daily on days 1-5. Treatment continues every 4 weeks for a maximum of 1 year in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive temozolomide as in arm I and whole brain radiotherapy on days 8-12 and 15-19 during the first course of chemotherapy.

Quality of life is assessed before beginning each course and then every 4 weeks after completion of study drug.

Patients are followed every 4 weeks.

PROJECTED ACCRUAL: A total of 250 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed unresectable metastatic melanoma

  * Must have asymptomatic brain metastasis that is not amenable to surgery or stereotactic radiosurgery (gamma knife, Linac)
  * Must have concurrent visceral/soft tissue metastases
* At least 1 site of measurable disease (not necessarily the brain metastasis)
* Documented evidence of disease progression defined by 1 of the following conditions:

  * More than 25% increase in the size of at least 1 measurable lesion
  * Appearance of a new lesion
  * A significant increase in the size of nonmeasurable disease
* No neurological symptoms, including signs of elevated intracranial pressure

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* SGOT or SGPT less than 3 times ULN
* Alkaline phosphatase less than 3 times ULN

Renal:

* Urea less than 1.5 times ULN
* Creatinine less than 1.5 times ULN

Other:

* No frequent vomiting or medical condition (e.g., partial bowel obstruction) that would interfere with oral medication intake
* No other prior or concurrent malignancy except surgically cured carcinoma in situ of the cervix or basal cell or squamous cell skin cancer
* No uncontrolled infection
* HIV negative
* No AIDS-related illness
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No psychological, familial, sociological, or geographical condition that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior cytokine via isolated limb perfusion for local-regional melanoma allowed
* No other prior cytokine for metastatic melanoma
* No concurrent colony-stimulating factors, including epoetin alfa or filgrastim (G-CSF)
* No other concurrent immunologic or biologic therapy

Chemotherapy:

* Prior chemotherapy via isolated limb perfusion for local-regional melanoma allowed
* No other prior chemotherapy for metastatic melanoma
* No other concurrent chemotherapy

Endocrine therapy:

* Concurrent corticosteroids allowed during radiotherapy (arm II only)
* No concurrent hormonal therapy

Radiotherapy:

* See Disease Characteristics
* No other concurrent radiotherapy

Surgery:

* See Disease Characteristics
* Recovered from the effects of any prior major surgery

Other:

* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2001-04; Primary Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juergen C. Becker, MD, PhD, Study Chair — Universitaets-Hautklinik Wuerzburg
Locations (33):
- Krankenhaus der Elisabethinen, Linz, Austria
- Belgium (4):
  - Institut Jules Bordet, Brussels
  - Hopital Universitaire Erasme, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Clinique Notre Dame de Grace, Gosselies
- Onkologicka Klinka A Onkologicka Lab, Prague, Czechia
- France (6):
  - CHU de Bordeaux - Hopital Pellegrin, Bordeaux
  - CHU Ambroise Pare, Boulogne-Billancourt
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Hopital L'Archet - 2, Nice
  - Centre Eugene Marquis, Rennes
  - Institut Gustave Roussy, Villejuif
- Germany (8):
  - Universitaetsklinikum Benjamin Franklin, Berlin
  - Federal Armed Forces Hospital of Ulm - Department of Dermatology, Blaustein
  - Universitaets - Augenklinik - Erlangen, Erlangen
  - Georg August Universitaet, Göttingen
  - Haematologisch-Onkologische Praxis Altona, Hamburg
  - III Medizinische Klinik Mannheim, Mannheim
  - Eberhard Karls Universitaet, Tübingen
  - Universitaet Wuerzburg/Hautkrankheiten, Würzburg
- Istituto Nazionale per la Ricerca sul Cancro, Genoa (Genova), Italy
- Netherlands (2):
  - University Medical Center Nijmegen, Nijmegen
  - Erasmus University Medical Center, Rotterdam
- Norwegian Radium Hospital, Oslo, Norway
- Instituto Portugues de Oncologia de Francisco Gentil - Centro de Lisboa, Lisbon, Portugal
- UniversitaetsSpital, Zurich, Switzerland
- United Kingdom (7):
  - Addenbrooke's NHS Trust, Cambridge, England
  - St. James's Hospital, Leeds, England
  - Royal Marsden NHS Trust, London, England
  - Christie Hospital N.H.S. Trust, Manchester, England
  - Weston Park Hospital, Manchester, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - Southend NHS Trust Hospital, Westcliff-on-Sea, England